CLINICAL TRIAL: NCT06971120
Title: CASI-Plus: A Mobile Health (mHealth) Tool for Client Engagement to Improve Ukraine's Assisted Partner Services (APS) Program Workflow and HIV Testing Outcomes (Aim 1)
Brief Title: CASI-Plus mHealth for Ukraine's APS Program (Aim 1)
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Nancy Puttkammer, Associate Professor, Global Health, University of Washington
Other Study IDs: STUDY00015808-Aim 1
Record Dates: First submitted 2025-04-23; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: HIV Infection
Keywords: Ukraine; HIV testing; partner notification
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Clients living with HIV: Clients living with HIV who participate in HIV index testing services
- Healthcare workers: Healthcare workers employed in primary care HIV clinics where HIV index testing services are provided

SUMMARY:
The CASI-Plus mHealth intervention seeks to improve partner elicitation and testing as part of assisted partner services (APS) in Ukraine, through a mHealth client engagement tool using computer-assisted self-interview (CASI). APS is a strategy for contact tracing and HIV testing for the high-risk sexual and needle-sharing partners of patients known to be living with HIV. This implementation science research will provide useful evidence on whether CASI-Plus can improve partner elicitation and HIV testing in a routine APS program operating at scale, toward the ultimate goal of linkage to HIV prevention and treatment services among those at highest risk of HIV. The aims are:

1. Aim 1 (R21): Conduct formative research from health worker and client perspectives to design the CASI-Plus mHealth intervention.
2. Aim 2 (R21): In a randomized controlled trial (RCT), assess adoption of CASI-Plus and its impact on contact elicitation. [NOTE: Aim 2 is covered under ClinicalTrials.gov record #NCT05826977]

Participants will integrate CASI-Plus as part of the APS services workflow to collect information from clients on sexual partners, needle-sharing partners, and biological children with risk of HIV exposure, and on self-reported partner notification and partner HIV testing outcomes.

The investigators will compare APS clients using CASI-Plus to APS clients receiving standard APS services, to see if the contact index (number of partners named per index client enrolled in APS services) and the HIV testing index (number of partners with unknown HIV status tested per index client enrolled in APS services) increase with use of CASI-Plus.

DETAILED DESCRIPTION:
In December 2016, the World Health Organization (WHO) recommended scale-up of assisted partner notification services (APS) as a strategy to increase HIV testing among persons living with HIV (PLWH). APS offers PLWH assistance to confidentially notify their sex and needle-sharing partners of their exposure and link them to testing and treatment. Randomized controlled trials (RCTs) have shown that APS increases HIV testing and case-finding, and is cost-effective. APS is scalable in routine practice, but typically with lower HIV case-finding than was observed in RCTs. APS outcomes are sub-optimal when recipients only name their current sex partner, or when partner notification and testing does not occur. There are an estimated 240,000 PLWH in Ukraine, of whom roughly three in four know their HIV status. While population-level HIV prevalence is 1.0%, prevalence among persons who inject drugs (PWID) and men who have sex with men (MSM) is 23% and 8%, respectively.

In 2019, the Ukraine Ministry of Health began scaling APS services. Despite trainings that emphasized the need to elicit >1 partner for each index client, health workers (HW) elicited only 1.14 for sexual and needle-sharing partners per index client, on average.16 Only 5.6% of APS clients identified as MSM or PWID and 45.9% of partners with unknown status had not yet completed HIV testing after 30 days.

The CASI-Plus mHealth intervention seeks to improve partner elicitation and testing, through a mHealth client engagement tool using computer-assisted self-interview (CASI). The CASI-Plus tool supports the initial APS encounter (providing information on how APS works, eliciting names of all sexual or injection partners, screening for risk of intimate partner violence [IPV], and planning for partner notification), and facilitates case management through partner testing (via repeat follow-up surveys to assess for barriers to notification, interest in provider assistance, IPV, and completion of notification). While CASI has reduced social desirability bias in surveys of sexual behavior across diverse settings, it has not yet been used in APS programs in low- or middle-income countries (LMICs). This implementation science research will provide useful evidence on whether CASI-Plus can improve partner elicitation and HIV testing in a routine APS program operating at scale, toward the ultimate goal of linkage to HIV prevention and treatment services among those at highest risk of HIV.

Aim 1 (R21): Conduct formative research from health worker and client perspectives to design the CASI-Plus mHealth intervention. Approach: The investigators will complete in-depth interviews with APS clients (N=10-15) and focus group discussions with HWs (N=3 groups of 8-15 HWs each) to elicit barriers to partner elicitation and testing, use this information to design the CASI-Plus tool and its integration within the APS workflow, and provide feedback on the tool's technical performance, usability, and acceptability. Hypothesis: CASI-Plus will be perceived by both clients and HWs as easy to navigate, acceptable, and technically sound.

ELIGIBILITY:
Inclusion Criteria for clients:

1. age 18 and over;
2. participated in APS services within the past 12 months at the study clinic;
3. willing to come to the clinic to participate in an in-depth interview about the intervention design; and
4. provide informed consent to participate in the study.

Inclusion Criteria for Health Workers:

1. age 18 and over;
2. employed at the study site;
3. have participated in delivery of HIV testing, prevention, care and/or treatment services at the health facility during the past year; and
4. provide informed consent to participate in the study.

Exclusion Criteria:

* Does not meet one or more inclusion criteria

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Clients are purposefully selected HIV index testing clients at one of the study sites (Chernihiv). Health workers are purposefully selected employees who are involved in delivering HIV index testing services at the two study sites (Chernihiv and Dnipro).
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2023-05-24 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Usability of CASI-Plus tool (client perspective) | Usability assessment will take place during months 1-12 (during development and testing of the CASI-Plus tool).
  The investigators will assess usability through qualitative interviews with clients.
Usability of CASI-Plus tool (health worker perspective) | Qualitative usability assessment will take place during months 1-12 (during development and testing of the CASI-Plus tool).
  The investigators will assess usability through qualitative interviews with healthcare workers.
Usability of CASI-Plus tool (health worker perspective) | Survey-based usability assessment will take place during the last 3 months of the study.
  The investigators will assess usability through surveys with healthcare workers. The survey includes adapted items from the System Usability Scale (SUS) which assesses dimensions of usability on a Likert scale, as well as customized, project specific items.

SECONDARY OUTCOMES:
Heuristic evaluation of CASI-Plus | Heuristic evaluation will take place in months 12-15 of the study.
  Health workers at the study sites and Ukrainian study team members will use a custom tool to document usability concerns based on common usability heuristics. The heuristic evaluation tool includes 16 heuristics applied to 12 sub-sections of the CASI-Plus tool. Users can document any issue that arises during prototype testing based on 5 test scripts (sample cases) as well as ad hoc testing. The can rate the severity of the issue identified (low, middle, high severity), and identify recommendations for fixing each issue.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Puttkammer, PhD, MPH, Principal Investigator — International Training and Education Center for Health, University of Washington
Locations (2):
- Ukraine (2):
  - Municipal Enterprise "Chernihiv Regional Hospital" of the Chernihiv Regional Council "Center for HIV/AIDS and Hepatitis Prevention", Chernihiv, Chernihiv Oblast
  - Municipal Enterprise "Dnipropetrovsk Regional Medical Center for Socially Significant Diseases" of the Dnipropetrovsk Regional Council, Dnipro, Dnipropetrovsk Oblast

IPD SHARING:
Plan to Share IPD: Yes
Shared individual participant data (IPD) will include IPD that underlie the results reported in published articles, after deidentification (text, tables, figures, and appendices). Anyone who wishes to access the data and who provides a methodologically sound proposal, may request access IPD. Researchers will be asked to submit a request in writing describing their qualifications including their certification by their local institutional review board (IRB), analytic plans and other uses of the data/resources, and plans to secure the confidentiality and safety of the data. They will be required to agree in writing that they will not share the data with others, will use it only for the research purpose(s) delineated, and will return or destroy the data upon completion. Proposals should be directed to Nancy Puttkammer (nputt@uw.edu). Given the sensitive nature of the data the investigators are collecting, including HIV diagnosis, the data will not be shared in a public access file.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Beginning 9 months and ending 36 months following article publication.